CLINICAL TRIAL: NCT01625169
Title: Antiretroviral Drug Concentrations and HIV Viral Load in Breast Milk and Plasma in HIV+ Women Receiving HAART (Highly Active Antiretroviral Therapy) Therapy: Etravirine (ETR) Pharmacokinetics (PK) in Breast Milk and Plasma
Brief Title: Etravirine Pharmacokinetics and HIV Viral Load in Breast Milk and Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Tibotec Therapeutics, a Division of Ortho Biotech Products, L.P., USA (Industry)
Responsible Party: Principal Investigator, LaShonda, Assistant Prof of Clinical Pediatrics, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HS-09-00698
Record Dates: First submitted 2012-06-12; First posted 2012-06-21 (Estimated); Results first posted 2014-08-07 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: HIV
Keywords: Pharmacokinetics; HIV; Breast milk
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HIV + pregnant women (Other): Etravirine pharmacokinetics in breast milk and plasma. Etravirine 200mg PO BID for 14 days with PK on days 5 and 14
  Interventions: Drug: Etravirine pharmacokinetics in breast milk and plasma

INTERVENTIONS:
Drug: Etravirine pharmacokinetics in breast milk and plasma — HIV+ pregnant women will receive etravirine 200mg PO BID for 14 days postpartum. PK will be done on postpartum days 5 and 14.

SUMMARY:
HIV positive pregnant women who receive potent combination antiretroviral therapy over at least the last trimester of pregnancy, and who have proper obstetric interventions and are able to avoid breast feeding, decrease the risk of having an infected infant to about 1%. Breast milk HIV-1 RNA (cell free) viral load is significantly associated with breast milk transmission, and a 2-fold increased risk of transmission associated with every 10-fold increase in breast milk viral load has been reported. In addition, cell associated virus (HIV DNA) was associated with a significant increase in risk of transmission independent of the level of cell-free viral RNA.

However, multiple studies of HIV positive women giving birth have shown that exclusive breast-feeding carries a much lower risk of HIV transmission than mixed breast-feeding (defined as breast milk along with complementary food, other milk, and/or infant formula). The proposed study will measure the antiretroviral (ARV) drug etravirine concentrations in blood and breast milk in postpartum HIV positive women on HAART therapy. The short-term goal is to determine how much etravirine penetrates into breast milk, and whether it leads to undetectable HIV viral load in the breast milk and therefore has the potential to decrease the risk of transmission of HIV through breast milk. The long term goal is to see if breast milk HIV levels can be lowered sufficiently to prevent maternal to child transmission (MTCT) of HIV in infants receiving only breast feeding in resource poor areas.

ELIGIBILITY:
Inclusion Criteria:

1. HIV+ pregnant women on HAART for the prevention of MTCT w/ undetectable viral load at time of delivery (w/i 30 days of delivery).
2. 18 years and older
3. Only women who are deemed by the physician as being capable of understanding that HIV positive women should not breastfeed will be approached.
4. Life expectancy greater than 6 months
5. No known allergies to etravirine
6. Willingness of subject to adhere to protocol requirements.

Exclusion Criteria:

1. Pregnant women with medical or psychological contraindications to breast milk expression.
2. Requirements for prohibited medications:

   * ARV: Tipranavir/ritonavir, fosamprenavir/ritonavir, atazanavir/ritonavir, and protease inhibitors administered without ritonavir, nonnucleoside reverse transcriptase inhibitor (NNRTIs).
   * Alternative/CAM: St. John's wort
   * Anticonvulsants: Phenobarbital, carbamazepine , phenytoin
   * Anti-infectives: Rifampin

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-04; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: LaShonda Y Spencer, MD, Principal Investigator — University of Southern California
Locations (1):
- LAC+USC MCA Clinic, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV + Pregnant Women: Etravirine PK on days 5 and 14
  Etravirine pharmacokinetics in breast milk and plasma: HIV+ pregnant women will receive etravirine for 14 days postpartum. PK will be done on postpartum days 5 and 14.
Period: Overall Study
Arm/Group | HIV + Pregnant Women
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- HIV + Pregnant Women: Etravirine PK on days 5 and 14
  Etravirine pharmacokinetics in breast milk and plasma: HIV+ pregnant women will receive etravirine for 14 days postpartum. PK will be done on postpartum days 5 and 14.
  There is only one arm- all pregnant women enrolled into the study will receive Etravirine 200mg PO bid for 14 days postpartum
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 9
Age, Continuous [Median (Full Range); unit: years] | 28.1 [21 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 9
Previous Pregnancies [Median (Full Range); unit: pregnancies]
  Gravida | 3 [1 to 8]
  Parity | 2 [0 to 6]
  Abortion | 1 [0 to 3]
Type of Delivery [Number; unit: participants]
  C-section | 2
  Vaginal | 7
Timing of Delivery [Number; unit: number participants]
  Term | 8
  Preterm | 1
Previous Breast Feeding [Number; unit: participants] — Data only available for 8 participants.
  participants
    Yes | 1
    No | 7
Absolute CD4 at Delivery [Median (Full Range); unit: cells/ml] | 437 [157 to 913]

OUTCOME MEASURES:

1. Primary Outcome: Peak Plasma Concentration of Etravirine in Plasma
Description: Cmax ng/ml
  Note: One participant did not complete the Day 5 evaluation.
Time Frame: Day 5
Population: Note: One participant did not complete the Day 5 evaluation.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng/ml | 497.6 (261.77)

2. Primary Outcome: Peak Concentration of Etravirine in Breast Milk
Description: Cmax ng/ml
  Note: One participant did not complete the Day 5 evaluation.
Time Frame: day 5
Population: Note: One participant did not complete the Day 5 evaluation.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng/ml | 685.4 (477.7)

3. Primary Outcome: Peak Concentration of Etravirine in Breast Milk
Description: Cmax ng/mL
Time Frame: day 14
Population: Note: One participant did not complete the Day 14 evaluation.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng/ml | 1805.4 (1390.0)

4. Primary Outcome: Peak Plasma Concentration of Etravirine in Plasma
Description: Cmax ng/mL
Time Frame: day 14
Population: Note: One participant did not complete the Day 14 evaluation.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng/ml | 564.6 (412.86)

5. Primary Outcome: Area Under the Curve (AUC) 0-12 for Plasma
Description: AUC 0-12 ng*hr/ml
Time Frame: Day 5: 0, 2,4, 8 and 24 hours post dose
Population: One participant did not complete Day 5 visit.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng*hr/ml | 3622.1 (2020.3)

6. Primary Outcome: Area Under the Curve (AUC) 0-12 for Plasma
Description: AUC 0-12 ng*hr/ml
Time Frame: Day 14: 0, 2,4, 8 and 24 hours post dose
Population: One participant did not complete D14 visit.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng*hr/ml | 4096 (2999.63)

7. Primary Outcome: Area Under the Curve (AUC) 0-12 for Breast Milk
Description: AUC 0-12 ng*hr/ml
Time Frame: Day 5
Population: One participant did not complete D5 visit.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng*hr/ml | 4371.9 (3491.8)

8. Primary Outcome: Area Under the Curve (AUC) 0-12 for Breast Milk
Description: AUC 0-12 ng*hr/ml
Time Frame: Day 14
Population: One participant did not complete D14 visit.
Measure: Mean (Standard Deviation); unit: ng*hr/ml
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
ng*hr/ml | 12953.7 (10200.4)

9. Secondary Outcome: HIV Viral Load in Breast Milk and Plasma
Description: Positive HIV RNA in breast milk and plasma- LDL 40 copies/ml
Time Frame: Day 5
Population: One participant did not complete Visit D5.
Measure: Number; unit: participants
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
participants
  Breast milk | 0
  Plasma | 1

10. Secondary Outcome: HIV Viral Load in Breast Milk and Plasma
Description: Positive HIV RNA in breast milk and plasma- LDL 40 copies/ml
Time Frame: Day 14
Population: One participant did not complete D14 visit.
Measure: Number; unit: participants
Arm/Group | HIV + Pregnant Women
Number analyzed (Participants) | 8
participants
  Breast milk | 2
  Plasma | 0

ADVERSE EVENTS:
Time Frame: Adverse Event reporting was collecting during the study and up through the last study visit.
Description: There were no significant toxicities or adverse events attributable to Etravirine administration in any of the subjects who received study drug. Safety labs were obtained at D14 visit. No lab toxicities were observed.
Arm/Group | HIV + Pregnant Women
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 6/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HIV + Pregnant Women (N=9)
Diarrhea (Gastrointestinal disorders) | 1 (1) — One patient out of 9 (11%) reported diarrhea at the D5 PK visit.
Headache (Nervous system disorders) | 1 (1) — 1 of 9 (11%) reported a self-resolving headache on D14; not likely to be related to ETR.
Breast Tenderness (Skin and subcutaneous tissue disorders) | 6 (6) — 66% of the subjects complained of breast tenderness related to pumping.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes